CLINICAL TRIAL: NCT05450952
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effects of a Theanine Formulation on Stress, Burnout, Mood, and Sleep in Individuals Who Report Occasional Moderate or High Levels of Stress
Brief Title: Evaluate the Effects of a Theanine Formulation on Stress, Burnout, Mood, and Sleep in Individuals Who Report Occasional Moderate or High Levels of Stress
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Electronic questionnaires not being completed in a timely manner
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol CL111
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Stress
Keywords: Burnout; Mood; Sleep; Fatigue
MeSH Terms: conditions — Burnout, Psychological; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Dietary Supplement (Theanine Formulation)
  Interventions: Dietary Supplement: Theanine Formulation
- Placebo (Placebo Comparator): Placebo Tablet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Theanine Formulation — Theanine Formulation Tablet
  Arms: Active
Dietary Supplement: Placebo — Placebo Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of the theanine formulation on stress, burnout, mood, and sleep in male and female subjects who are generally healthy

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study to evaluate the effects of a theanine formulation on stress, burnout, mood, and sleep in individuals who are generally healthy.

Participants will be asked to completed assessments and questionnaires as well as obtain a self saliva sample.

The primary objective is to evaluate the change in response to the theanine formulation on stress from completed questionnaires at Day 1, Day 7 and Day 28 relative to the baseline values. The questionnaires utilized for this objective include Depression, Anxiety and Stress Scale (DASS-21), State-Trait Anxiety Inventory (STAI) and Perceived Stress Scale (PSS-14).

The secondary objective is to evaluate the change in response to the theanine formulation on burnout, mood, and sleep at Day 1, Day 7 and Day 28 relative to the baseline values. The questionnaires assessments utilized for this objective include Leeds Sleep Evaluation Questionnaires (LSEQ), Maslach Burnout Inventory General Survey (MBI-GS), Visual Analog Mood Scale (VAMS), Short Form-36 Health Survey (SF-36) and Cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, 21-65 years of age
2. A BMI of 18.5-34.9
3. Admits to having occasional periods of moderate or severe stress
4. Indicating a DASS score > 19 (identification as having moderate, severe, or extremely severe stress)
5. Indicating a PSS-14 score > 19 (identification as having moderate or high perceived stress)
6. Have personal access to and able to operate a smartphone, tablet, or computer with enough memory to accommodate additional application(s) and have a reliable internet service
7. Able to print out and return documents by email (preferred)or mail
8. If have a history of testing positive for coronavirus SARS-CoV2 (COVID-19, being asymptomatic for a minimum of 14 days and have a negative COVID-19 antigen test
9. Able to take saliva specimens with a swab and store them immediately in a freezer before breakfast, lunch, dinner, and bedtime on four different days during the study
10. Generally healthy and having no difficulty swallowing a tablet
11. Have sufficient freezer space to hold a minimum of 2 saliva test kits (approximately the size of 2 ice cream cartons)
12. Has regular daytime work hours or shifts, if employed (regular shift excludes night shift workers and those with rotating shifts)
13. Has been generally weight stable for the past six months (+/- 6 lbs.)
14. Willing and able to give written informed consent
15. Clearly understands the procedures and study requirements
16. Willing and able to comply with all study procedures, including following recommendations to maintain their usual diet and regular activity, as per protocol
17. Able to communicate, including reading, in English
18. Has not taken any nutritional supplements that may contain any of the active component of the study product including L-theanine for a minimum of 14 days before Screening/baseline and for the duration of the study period

Exclusion Criteria:

1. Not having the basic skills needed to operate a smartphone, tablet, or computer
2. Unwilling to limit daily caffeine intake to less than 400 mg caffeine per day (~ 95 mg caffeine in a cup of regular coffee) and refrain from consuming any caffeinated beverages/foods after 2 PM daily for the duration of the study
3. Having smoked any cigarette, electronic cigarette, cigar, pipe, or used a recreational drug as well as any product containing cannabidiol (CBD) or tetrahydrocannabinol (THC) in the past 30 days prior to Screening/baseline
4. Having donated blood within 30 days before Screening/baseline
5. Having been diagnosed with dysphagia or difficulty swallowing
6. Having participated in another study within 30 days prior to Screening/baseline
7. Being pregnant or planning on becoming pregnant during study participation; or breast feeding
8. History of allergy or sensitivity to any component of the study products including L-theanine, microcrystalline cellulose, hydroxypropyl methylcellulose, stearic acid, silica, silicon dioxide, vegetable stearate, croscarmellose sodium or glycerin
9. Are not participating in a stress management program and will not for the duration of the study participation.
10. Unable to avoid any form of intense exercise or a significant change in your exercise routine during the day of saliva specimen collection
11. Currently taking supplements including melatonin, 5-hydroxytryptophan, Calamus, California poppy, St. John's wort, S-adenosylmethionine (SAM-E), catnip, hops, kava, valerian, Jamaican dogwood, skullcap, yerba mansa, Hawaiian baby woodrose, L-theanine, magnesium, or any other supplement for stress, burnout, mood, or sleep. These may preclude participation in the study dependent the judgment of the Study Investigator/Sub-Investigator
12. Having been diagnosed, received medical treatment, taking medication/supplements daily for the following medical condition(s):

    * Stress disorder (including post-traumatic stress disorder [PTSD])
    * Sleep disorder (including insomnia diagnosed by a physician)
    * Psychiatric disorder (bipolar disorder, manic disorder, schizophrenia, apathetic [inherited] disorder), that include antidepressant drugs, including selective serotonin reuptake inhibitors (SSRIs), tricyclic and atypical antidepressants; benzodiazepines; phenothiazines, central nervous system (CNS) depressants as well as the following medications: dextromethorphan, meperidine, monoamine oxidase inhibitors (MAOIs), pentazocine and tramadol. These may preclude participation in the study dependent on the judgment of the Study Investigator/Sub-Investigator.
    * Acute or chronic inflammatory or autoimmune disease (including rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis, Sjögren's syndrome, polymyalgia rheumatica, inflammatory bowel disease, psoriatic arthritis, fibromyalgia, or chronic fatigue syndrome)
    * Active infection
    * Active periodontal disease
13. Presence of active or recurring clinically significant conditions as follows:

    * Diabetes mellitus (except on a stable dose of Metformin up to 1000 mg per day only for managing the diabetes mellitus for > 3 months before Screening/baseline, unlikely to change medication or dose during the study, and under the care of a physician having seen the physician within 6 months before Screening/baseline)
    * Endocrine disease (other than diabetes mellitus)
    * Eating disorder
    * Cardiovascular disease including heart and blood vessel disease, arrhythmia, heart attack, stroke, or heart valve problem
    * Gastrointestinal disease including gallbladder problems, gallstones, or biliary tract obstruction
    * Thyroid disease (except on a stable dose of medication for ≥ 3 months before Screening/baseline and unlikely to change medication or dose during the study)
    * Hypertension (except on a stable dose of medication for ≥ 3 months before Screening/baseline and unlikely to change medication or dose during the study)
    * Neurologic condition/disease
    * Cancer (including skin cancer) which has been treated ≥ 5 years before Screening/baseline or at the discretion of the Study Investigator/Sub-Investigator
    * Liver, pancreatic, and kidney disease
    * Pulmonary disease
    * Blood coagulation disorder or other hematologic disease
    * Any other condition or medication that may preclude study participation in the judgement of the Study Investigator/Sub-Investigator
14. Currently taking or having taken within the 30 days before Screening/baseline any hormone replacement therapy (including dehydroepiandrosterone (DHEA), estrogen, progesterone, or testosterone), except those utilized as a method of birth control and which have been taken for > 3 months with no anticipated change for the duration of the study period
15. Having had a surgical procedure or having an internal medical device which, in the judgment of the Study Investigator/Sub-Investigator, would preclude participation in the study
16. Currently consumes more than 4 standard alcoholic drinks per week for women and 7 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
17. Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges, and tangelos for the duration of the study period
18. History of known or suspected substance abuse (e.g., alcohol, opiates, benzodiazepines, or amphetamines)
19. Having any other circumstance that may preclude study participation in the judgment of the Study Investigator/Sub-Investigator, including use of other nutritional supplements, which will be evaluated on a case-by-case basis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale-21 (DASS-21) | 28 days
  Assessment of the mean change in the results of Depression, Anxiety and Stress Scale-21 (DASS-21) from baseline. There are 21 items consisting of three scales (Depression, Anxiety and Stress) contains 7 items and scores from each scale can range from 0-56. The lower the scores for each scale indicates a better outcome.
State-Trait Anxiety Inventory (STAI) | 28 days
  Assessment of the mean change in the results of the State-Trait Anxiety Inventory (STAI) from baseline. This is a 20-item questionnaire which includes separate measures of state and trait anxiety. The total scores range from 0-63. The lower the score indicates a better outcome.
Perceived Stress Scale (PSS-14) | 28 days
  Assessment of the mean change in the results of the Perceived Stress Scale (PSS-14) from baseline. There are 14 items and total scores range from 0-56. The lower the score indicates a lower level of stress.

SECONDARY OUTCOMES:
Leeds Sleep Evaluation Questionnaire (LSEQ) | 28 days
  Assessment of the mean change in the results of the Leeds Sleep Evaluation Questionnaires (LSEQ) from baseline. This questionnaire consists of ten self-rating questions related to four consecutive aspects of sleep (getting to sleep, quality of sleep, awakening from sleep and behavior following sleep). The total LSEQ score can range from 0-100. The higher the total global LSEQ score indicates a better outcome.
Maslach Burnout Inventory (MBI-GS) | 28 days
  Assessment of the mean change in the results of Maslach Burnout Inventory (MBI-GS) from baseline. This survey consists of 16 statements of job-related feelings. It consists of 3 subscales including Emotional Exhaustion, Depersonalization and Professional Accomplishment. The total score can range from 0 to 96. The lower the score for the Emotional Exhaustion and Depersonalization components represent a better outcome and a higher score for the Professional Accomplishment represents a better outcome.
Visual Analog Mood Scales (VAMS) | 28 days
  Assessment of the mean change in the results of Visual Analog Mood Scales (VAMS) from baseline. These scales measure eight mood states including Afraid, Confused, Sad, Angry, Energetic, Tired, Happy and Tense. Each score for each mood ranges from 0 to 100. The lower the score for each mood represents a minimal level of that mood and the higher score represents the greater level of that mood.
Short Form -36 Health Survey (SF-36) | 28 days
  Assessment of the mean change in the results of the Short Form-36 Health Survey (SF-36) from baseline. This is a 36-item questionnaire that covers eight domains including physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue and general health perceptions. The scores from each domain can range from 0 to 100. The higher the scores for each domain indicates a better outcome.
Cortisol Levels | 28 days
  Assessment of the mean change in the results of Cortisol levels from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn RS, Lee YJ, Choi JY, Kwon HB, Chun SI. Salivary cortisol and DHEA levels in the Korean population: age-related differences, diurnal rhythm, and correlations with serum levels. Yonsei Med J. 2007 Jun 30;48(3):379-88. doi: 10.3349/ymj.2007.48.3.379. PMID 17594144
- [Background] Borzelleca JF, Peters D, Hall W. A 13-week dietary toxicity and toxicokinetic study with l-theanine in rats. Food Chem Toxicol. 2006 Jul;44(7):1158-66. doi: 10.1016/j.fct.2006.03.014. Epub 2006 Apr 26. PMID 16759779
- [Background] Dallal, G. (2021). www.Randomization.com. Retrieved from http://www.randomization.com
- [Background] Drugs, O. o. N. (2005). Guidance for Industry. Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. Retrieved from https://www.fda.gov/media/72309/download
- [Background] Fernandez-Guasti A, Fiedler JL, Herrera L, Handa RJ. Sex, stress, and mood disorders: at the intersection of adrenal and gonadal hormones. Horm Metab Res. 2012 Jul;44(8):607-18. doi: 10.1055/s-0032-1312592. Epub 2012 May 11. PMID 22581646
- [Background] Hidese S, Ogawa S, Ota M, Ishida I, Yasukawa Z, Ozeki M, Kunugi H. Effects of L-Theanine Administration on Stress-Related Symptoms and Cognitive Functions in Healthy Adults: A Randomized Controlled Trial. Nutrients. 2019 Oct 3;11(10):2362. doi: 10.3390/nu11102362. PMID 31623400
- [Background] Hidese S, Ota M, Wakabayashi C, Noda T, Ozawa H, Okubo T, Kunugi H. Effects of chronic l-theanine administration in patients with major depressive disorder: an open-label study. Acta Neuropsychiatr. 2017 Apr;29(2):72-79. doi: 10.1017/neu.2016.33. Epub 2016 Jul 11. PMID 27396868
- [Background] Higashiyama, A., Htay, H, Ozeki, M Et Al. (2011). Effects of L-theanine on attention and reaction time response. Journal of Functional Foods, 3, 171-178.
- [Background] Kakuda T, Hinoi E, Abe A, Nozawa A, Ogura M, Yoneda Y. Theanine, an ingredient of green tea, inhibits [3H]glutamine transport in neurons and astroglia in rat brain. J Neurosci Res. 2008 Jun;86(8):1846-56. doi: 10.1002/jnr.21637. PMID 18293419
- [Background] Kim EJ, Dimsdale JE. The effect of psychosocial stress on sleep: a review of polysomnographic evidence. Behav Sleep Med. 2007;5(4):256-78. doi: 10.1080/15402000701557383. PMID 17937582
- [Background] Kim S, Jo K, Hong KB, Han SH, Suh HJ. GABA and l-theanine mixture decreases sleep latency and improves NREM sleep. Pharm Biol. 2019 Dec;57(1):65-73. doi: 10.1080/13880209.2018.1557698. PMID 30707852
- [Background] Kimura K, Ozeki M, Juneja LR, Ohira H. L-Theanine reduces psychological and physiological stress responses. Biol Psychol. 2007 Jan;74(1):39-45. doi: 10.1016/j.biopsycho.2006.06.006. Epub 2006 Aug 22. PMID 16930802
- [Background] Levine A, Zagoory-Sharon O, Feldman R, Lewis JG, Weller A. Measuring cortisol in human psychobiological studies. Physiol Behav. 2007 Jan 30;90(1):43-53. doi: 10.1016/j.physbeh.2006.08.025. Epub 2006 Oct 19. PMID 17055006
- [Background] Lopes Sakamoto F, Metzker Pereira Ribeiro R, Amador Bueno A, Oliveira Santos H. Psychotropic effects of L-theanine and its clinical properties: From the management of anxiety and stress to a potential use in schizophrenia. Pharmacol Res. 2019 Sep;147:104395. doi: 10.1016/j.phrs.2019.104395. Epub 2019 Aug 11. PMID 31412272
- [Background] Miodownik C, Maayan R, Ratner Y, Lerner V, Pintov L, Mar M, Weizman A, Ritsner MS. Serum levels of brain-derived neurotrophic factor and cortisol to sulfate of dehydroepiandrosterone molar ratio associated with clinical response to L-theanine as augmentation of antipsychotic therapy in schizophrenia and schizoaffective disorder patients. Clin Neuropharmacol. 2011 Jul-Aug;34(4):155-60. doi: 10.1097/WNF.0b013e318220d8c6. PMID 21617527
- [Background] Nathan PJ, Lu K, Gray M, Oliver C. The neuropharmacology of L-theanine(N-ethyl-L-glutamine): a possible neuroprotective and cognitive enhancing agent. J Herb Pharmacother. 2006;6(2):21-30. PMID 17182482
- [Background] Perez-Valdecantos D, Caballero-Garcia A, Del Castillo-Sanz T, Bello HJ, Roche E, Cordova A. Stress Salivary Biomarkers Variation during the Work Day in Emergencies in Healthcare Professionals. Int J Environ Res Public Health. 2021 Apr 9;18(8):3937. doi: 10.3390/ijerph18083937. PMID 33918537
- [Background] Ritsner MS, Miodownik C, Ratner Y, Shleifer T, Mar M, Pintov L, Lerner V. L-theanine relieves positive, activation, and anxiety symptoms in patients with schizophrenia and schizoaffective disorder: an 8-week, randomized, double-blind, placebo-controlled, 2-center study. J Clin Psychiatry. 2011 Jan;72(1):34-42. doi: 10.4088/JCP.09m05324gre. Epub 2010 Nov 30. PMID 21208586
- [Background] Rogers PJ, Smith JE, Heatherley SV, Pleydell-Pearce CW. Time for tea: mood, blood pressure and cognitive performance effects of caffeine and theanine administered alone and together. Psychopharmacology (Berl). 2008 Jan;195(4):569-77. doi: 10.1007/s00213-007-0938-1. Epub 2007 Sep 23. PMID 17891480
- [Background] Rosner, B. (2006). Hypothesis Testing Two-Sample Inference. In Fundamentals of Biostatistics (6th ed., pp. 331-334): Duxbury Press.
- [Background] Sanford LD, Suchecki D, Meerlo P. Stress, arousal, and sleep. Curr Top Behav Neurosci. 2015;25:379-410. doi: 10.1007/7854_2014_314. PMID 24852799
- [Background] Scheid L, Ellinger S, Alteheld B, Herholz H, Ellinger J, Henn T, Helfrich HP, Stehle P. Kinetics of L-theanine uptake and metabolism in healthy participants are comparable after ingestion of L-theanine via capsules and green tea. J Nutr. 2012 Dec;142(12):2091-6. doi: 10.3945/jn.112.166371. Epub 2012 Oct 24. PMID 23096008
- [Background] Silva BKR, Quaresma FRP, Maciel EDS, Figueiredo FWDS, Sarraf JS, Adami F. Correlation Between Stress and Quality of Life Experienced by Caregivers: Perception of a Group of Healthcare Professionals. Open Nurs J. 2017 Sep 27;11:135-141. doi: 10.2174/1874434601711010135. eCollection 2017. PMID 29238419
- [Background] Tsujita S, Morimoto K. Secretory IgA in saliva can be a useful stress marker. Environ Health Prev Med. 1999 Apr;4(1):1-8. doi: 10.1007/BF02931243. PMID 21432164
- [Background] Unno K, Tanida N, Ishii N, Yamamoto H, Iguchi K, Hoshino M, Takeda A, Ozawa H, Ohkubo T, Juneja LR, Yamada H. Anti-stress effect of theanine on students during pharmacy practice: positive correlation among salivary alpha-amylase activity, trait anxiety and subjective stress. Pharmacol Biochem Behav. 2013 Oct;111:128-35. doi: 10.1016/j.pbb.2013.09.004. Epub 2013 Sep 16. PMID 24051231
- [Background] Weitzman ED, Fukushima D, Nogeire C, Roffwarg H, Gallagher TF, Hellman L. Twenty-four hour pattern of the episodic secretion of cortisol in normal subjects. J Clin Endocrinol Metab. 1971 Jul;33(1):14-22. doi: 10.1210/jcem-33-1-14. No abstract available. PMID 4326799
- [Background] WHO (2019) Burn out an occupation phenomenon. International Classification of Diseases. Retrieved from https://www.who.int/news/item/28-05-2019-burn-out-an-occupational-phenomenon-international-classification-of-diseases
- [Background] Williams JL, Everett JM, D'Cunha NM, Sergi D, Georgousopoulou EN, Keegan RJ, McKune AJ, Mellor DD, Anstice N, Naumovski N. The Effects of Green Tea Amino Acid L-Theanine Consumption on the Ability to Manage Stress and Anxiety Levels: a Systematic Review. Plant Foods Hum Nutr. 2020 Mar;75(1):12-23. doi: 10.1007/s11130-019-00771-5. PMID 31758301
- [Background] Yaribeygi H, Panahi Y, Sahraei H, Johnston TP, Sahebkar A. The impact of stress on body function: A review. EXCLI J. 2017 Jul 21;16:1057-1072. doi: 10.17179/excli2017-480. eCollection 2017. PMID 28900385
- [Background] Care, I. f. Q. a. E. i. H. (2020). Depression: What is burnout? Retrieved from https://www.ncbi.nlm.nih.gov/books/NBK279286/